CLINICAL TRIAL: NCT00761358
Title: To Verify the Efficacy of Z-338 in Subjects With Functional Dyspepsia, Focusing on the Assessment of Subjective Symptoms
Brief Title: To Verify the Efficacy of Z-338 in Subjects With Functional Dyspepsia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zeria Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 99010301
Record Dates: First submitted 2008-09-25; First posted 2008-09-29 (Estimated); Last update posted 2010-11-23 (Estimated); Status verified 2010-11

CONDITIONS: Functional Dyspepsia
Keywords: Acotiamide
MeSH Terms: interventions — Z 338

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Z-338 (Experimental)
  Interventions: Drug: Z-338
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Z-338 — Oral
  Arms: Z-338
Drug: Placebo — Oral
  Arms: placebo

SUMMARY:
The purpose of this study is to verify the superior efficacy of Z-338 to placebo in subjects with Functional Dyspepsia, focusing on the assessment of subjective symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Subjects showing at least one of the 4 symptoms (upper abdominal pain, upper abdominal discomfort, epigastric pain, epigastric burning) for at least 6 months before obtaining informed consent
* Subjects showing two or more of the following symptoms: upper abdominal pain, upper abdominal discomfort, post-prandial fullness, upper abdominal bloating, early satiety, nausea, vomiting and/or excessive belching for at least 3 months (one of them should be post-prandial fullness or early satiation)
* Bothersome symptoms should be post-prandial fullness, upper abdominal bloating or early satiety at the time of obtaining informed consent

Exclusion Criteria:

* Subjects with structural disease that is likely to explain the symptom (e.g., GERD, erosion, ulcer, hiatal hernia, bleeding, malignancy or Barrett's esophagus) confirmed by upper endoscopy at the obtaining informed consent
* Subjects have heartburn in last 12 weeks before obtaining informed consent
* Subjects with irritable bowel disease (IBS)
* Subjects with diabetes mellitus requiring treatment
* Subjects with serious anxiety disorder
* Subjects with depression and/or sleep disorder
* Subjects with biliary tract disease and/or pancreatitis (including chronic pancreatitis)

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 820 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-06 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
General impression at last visit in treatment period | 4 week
Elimination rate of post-prandial fullness, upper abdominal bloating and early satiety at last visit in treatment period | 4 week

SECONDARY OUTCOMES:
Individual symptom score | Every week
SF-NDI | At 0, 4 week and 4 week after treatment
General Impression | Every week
Laboratory tests | At 0, 4 week and 4 week after treatment
Adverse Event | 4 week treatment period and 4 week after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michio Hongo, Professor, Study Director — Tohoku University Hospital
Locations (2):
- Japan (2):
  - Hokkaido
  - Tokyo

REFERENCES:
- [Derived] Matsueda K, Hongo M, Tack J, Saito Y, Kato H. A placebo-controlled trial of acotiamide for meal-related symptoms of functional dyspepsia. Gut. 2012 Jun;61(6):821-8. doi: 10.1136/gutjnl-2011-301454. Epub 2011 Dec 9. PMID 22157329